CLINICAL TRIAL: NCT07215559
Title: A Phase 2, Parallel-Group, Double-Blind, Placebo-Controlled Study to Investigate Weight Reduction With Macupatide and Eloralintide, Alone or in Combination, in Adult Participants With Obesity or Overweight and With Type 2 Diabetes
Brief Title: A Study of Macupatide (LY3532226) and Eloralintide (LY3841136), Alone or in Combination, in Adults With Obesity or Overweight and With Type 2 Diabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27721; J2V-MC-GZLF (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-09; First posted 2025-10-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight; Diabetes Mellitus, Type 2
Keywords: GIP; Amylin
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Macupatide (Macupatide + Eloralintide Placebo) (Experimental): Participants will be administered macupatide subcutaneously (SC) and eloralintide placebo SC
  Interventions: Drug: Macupatide; Drug: Eloralintide Placebo
- Eloralintide (Elorlintide + Macupatide Placebo) (Experimental): Participants will be administered eloralintide SC and macupatide placebo SC
  Interventions: Drug: Eloralintide; Drug: Macupatide Placebo
- Macupatide + Eloralintide (Experimental): Participants will be administered eloralintide SC and macupatide SC
  Interventions: Drug: Macupatide; Drug: Eloralintide
- Placebo (Macupatide Placebo + Elorlintide Placebo) (Placebo Comparator): Participants will be administered eloralintide placebo SC and macupatide placebo SC
  Interventions: Drug: Macupatide Placebo; Drug: Eloralintide Placebo

INTERVENTIONS:
Drug: Macupatide — Administered SC
  Other Names: LY3532226
  Arms: Macupatide (Macupatide + Eloralintide Placebo); Macupatide + Eloralintide
Drug: Eloralintide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide (Elorlintide + Macupatide Placebo); Macupatide + Eloralintide
Drug: Macupatide Placebo — Administered SC
  Arms: Eloralintide (Elorlintide + Macupatide Placebo); Placebo (Macupatide Placebo + Elorlintide Placebo)
Drug: Eloralintide Placebo — Administered SC
  Arms: Macupatide (Macupatide + Eloralintide Placebo); Placebo (Macupatide Placebo + Elorlintide Placebo)

SUMMARY:
The purpose of this study is to investigate weight reduction with macupatide and eloralintide, alone or in combination, in adult participants with obesity or overweight and with type 2 diabetes. Participation in the study will last about 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Have an HbA1c ≥7.5% to ≤10.5% at screening
* Have been treated with any of the following, alone or in combination, for at least 3 months prior to screening

  * Diet and exercise
  * Stable dose of metformin
  * Sodium-glucose cotransporter-2 (SGLT2) inhibitor
* Have had a stable body weight (<5% body weight gain and/or loss) for the 3 months prior to screening
* Have a BMI of 27 or greater at screening

Exclusion Criteria:

* Have any form of diabetes other than type 2 diabetes
* Have a prior or planned surgical treatment for obesity, except prior liposuction or abdominoplasty, if performed >1 year prior to screening
* Have any of the following cardiovascular conditions within 3 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years, exceptions include

  * basal or squamous cell skin cancer
  * in situ carcinomas of the cervix, or
  * in situ prostate cancer
* Have been prescribed any of the following receptor agonists (RA) or their combination for any indication within the last 6 months:

  * amylin RA
  * dual amylin and calcitonin RA
  * glucagon-like peptide-1 receptor (GLP-1) RA
  * glucose-dependent insulinotropic peptide (GIP)/GLP-1 RA
  * GLP-1/glucagon (GCG) RAs, or
  * GIP/GLP-1/GCG RAs
* Have used excluded antihyperglycemic medications within 3 months prior to screening (including, but not limited to, sulfonylureas, dipeptidyl peptidase-4 inhibitors, alpha-glucosidase inhibitors, thiazolidinediones, and meglitinides
* Have used insulin for diabetic control within the prior year (short term use in certain situations allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 32

SECONDARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 32
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 32
Change from Baseline in Fasting Glucose | Baseline, Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (38):
- United States (22):
  - Prime Medical Group, LLC dba Gilbert Center for Family Medicine, LLC, Gilbert, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Pima Heart, Tucson, Arizona
  - SKY Clinical Research Network Group-Brown, Atlanta, Georgia
  - Teak Research Consults, Lawrenceville, Georgia
  - AGILE Clinical Research Trials, LLC, Sandy Springs, Georgia
  - Pivotal Research Solutions, Stonecrest, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Vector Clinical Trials, Las Vegas, Nevada
  - Premier Research, Trenton, New Jersey
  - Mercy Family Clinic, Dallas, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Aavon Clinical Trials, Richmond, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Kalo Clinical Research, West Valley City, Utah
  - Eastern Virginia Medical School (EVMS) Medical Group, Norfolk, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Universal Research Group, Tacoma, Washington
- Argentina (6):
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - CENUDIAB, Buenos Aires
  - CEDIC, CABA
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Go Centro Medico San Nicolás, San Nicolás
- Australia (8):
  - Emeritus Research, Botany
  - Core Research Group, Brisbane
  - Emeritus Research, Camberwell
  - Cornerstone Dermatology, Coorparoo
  - Momentum Darlinghurst, Darlinghurst, Sydney
  - CDH Research Institute Pty Ltd, Maroochydore
  - Momentum Sunshine, Melbourne
  - AIM Research, Merewether
- Puerto Rico (2):
  - San Juan Bautista School of Medicine - Clinical Research Unit, Caguas
  - Mgcendo Llc, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Macupatide (LY3532226) and Eloralintide (LY3841136), Alone or in Combination, in Adults With Obesity or Overweight and With Type 2 Diabetes — https://trials.lilly.com/en-US/trial/659876